CLINICAL TRIAL: NCT04794803
Title: Study on the Efficacy and Safety of Reparixin in the Treatment of Hospitalized Patients With COVID-19 Pneumonia
Brief Title: Reparixin in COVID-19 Pneumonia - Efficacy and Safety
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The sponsor has decided to start with a separate protocol for phase 3 and therefore this study was terminated with only phase 2.
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REPAVID-19; 2020-001645-40 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Results first posted 2022-03-17 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2022-05

CONDITIONS: Severe Pneumonia
Keywords: COVID-19
MeSH Terms: conditions — Pneumonia; COVID-19 | interventions — reparixin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reparixin (Experimental): Reparixin oral tablets 1200 mg TID for 7 days
  Interventions: Drug: Reparixin
- Standard of care (Active Comparator): Standard of care
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Reparixin — Reparixin was administered via oral tablets 1200 mg TID for 7 days. In case of improvement, treatment can be prolonged at discretion of the investigator up to a maximum of 21 days of treatment in total or live discharge from the hospital, whichever comes first.
  Other Names: Repertaxin L-lysine salt
  Arms: Reparixin
Drug: Standard of care — Standard of care
  Other Names: Control
  Arms: Standard of care

SUMMARY:
* Phase 2 Study Objectives: efficacy and safety of of Reparixin treatment as compared to the control arm in adult patients with severe COVID-19 pneumonia
* Phase 3 Study Objectives: efficacy and safety of Reparixin treatment as compared to the control arm in adult patients with moderate or severe COVID-19 pneumonia

DETAILED DESCRIPTION:
This clinical trial is an adaptive phase 2/3, randomized, controlled multicenter study on the efficacy and safety of Reparixin in the treatment of hospitalized patients with COVID-19 pneumonia. 48 patients are planned to be enrolled in Phase 2 and an estimated total of 111 patients are planned to be enrolled up to the end of Phase 3, with a randomization 2:1 Reparixin vs Control (Standard of care).

In the phase 2 segment of this study, patients are randomized 2:1 to Reparixin oral tablets 1200 mg (Group 1, active treatment) or standard of care (Group 2, control arm). In case of worsening (e.g. need of ICU and/or mechanical ventilation) after the first 24hrs, patients are offered a rescue medication with no restriction from the sponsor and fully based on their physicians' judgement.

In the phase 3 segment of this study, it is planned that patients are randomized 2:1 to Reparixin or standard of care. The Phase 3 design will be reassessed and decided based on the results of the Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Phase 2 Inclusion Criteria:

  1. Age 18 to 90.
  2. Confirmed COVID-19 diagnosis
  3. At least one of the following: # Respiratory distress, RR ≥ 30 breaths/min without oxygen; # Partial arterial oxygen pressure (PaO2) / Fraction of inspiration O2 (FiO2) >100 <300mmHg

  (1mmHg = 0.133kPa). 4. Chest imaging confirms lung involvement and inflammation. 5. Inflammatory status as documented by at least one of the following: Lactate dehydrogenase (LDH) > normal range, C-reactive protein (CRP) ≥ 100mg/L or IL-6 ≥ 40pg/mL, serum ferritin ≥ 900ng/mL, XDP >20mcg/mL.
* Phase 3 Inclusion Criteria: Same as above; other criteria TBD based on Phase 2 outcomes.

Exclusion Criteria:

• Phase 2/3 Exclusion Criteria:

1. Cannot obtain informed consent.
2. Severe hepatic dysfunction (Child Pugh score ≥ C, or AST> 5 times the upper limit); Severe renal dysfunction (estimated glomerular filtration rate ≤ 30mL / min / 1.73 m2) or receive continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
3. Patients with hypersensitivity to ibuprofen or to more than one non steroidal anti-inflammatory drug or to more than one medication belonging to the class of sulfonamides (e.g. sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib; hypersensitivity to sulphanilamide antibiotics alone, e.g. sulfamethoxazole, does not qualify for exclusion)
4. Severe, active bleeding such as hemoptysis, gastrointestinal bleeding, central nervous system bleeding, and nosebleeds within 1 month before enrollment.
5. Pregnant and lactating women and those planning to get pregnant.
6. Participated in other interventional clinical trials with investigational medicinal products, not considered suitable for this study by the researchers.
7. At the time of enrollment, patients not in a clinical condition compatible with the oral administration of the study drug.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD PhD, Principal Investigator — Ospedale San Raffaele; Alberto Zangrillo, MD PhD, Principal Investigator — Ospedale San Raffaele
Locations (4):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina de São Paulo, São Paulo, Brazil
- Italy (3):
  - Ospedale San Paolo, Milan, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Ospedale di Varese, Varese, Lombardy

REFERENCES:
- [Derived] Landoni G, Piemonti L, Monforte AD, Grossi P, Zangrillo A, Bucci E, Allegretti M, Goisis G, Gavioli EM, Patel N, De Pizzol M, Pasedis G, Mantelli F. A Multicenter Phase 2 Randomized Controlled Study on the Efficacy and Safety of Reparixin in the Treatment of Hospitalized Patients with COVID-19 Pneumonia. Infect Dis Ther. 2022 Aug;11(4):1559-1574. doi: 10.1007/s40121-022-00644-6. Epub 2022 May 26. PMID 35618953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 patients were screened and all of them were randomized to the assigned treatment group: 37 patients were randomised to receive Reparixin and 19 patients were randomised to receive standard of care.
Period: Overall Study
Arm/Group | Reparixin | Standard of Care
Started | 37 | 19
FAS Population | 36 | 19
Safety Set | 36 | 19
Per Protocol Set | 17 | 11
Completed | 27 | 11
Not Completed | 10 | 8
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Patient transferred to another centre for oxygen rehabilitation | 4 | 1
Not completed — Refused to continue the treatment | 1 | 0
Not completed — Patient admitted to ICU | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP. The FAS population was analyzed according to intention to treat (ITT) principle, i.e. by treatment allocation regardless the occurrence of intercurrent events.
Groups:
- Reparixin (FAS): Reparixin oral tablets 1200 mg TID for 7 days
  Reparixin: Reparixin was administered via oral tablets 1200 mg TID for 7 days. In case of improvement, treatment can be prolonged at discretion of the investigator up to a maximum of 21 days of treatment in total or live discharge from the hospital, whichever comes first.
- Standard of Care (FAS): Standard of care
  Standard of care: Standard of care
- Total: Total of all reporting groups
Arm/Group | Reparixin (FAS) | Standard of Care (FAS) | Total
Number analyzed (Participants) | 36 | 19 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 11 | 33
  >=65 years | 14 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (13.5) | 63.6 (14.2) | 61.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 26 | 16 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic Or Latino | 18 | 8 | 26
  Not reported | 3 | 1 | 4
  Unknown | 11 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 32 | 16 | 48
  Black Or African American | 1 | 1 | 2
  Brown | 3 | 1 | 4
  Other Ethnic Group | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 2 | 2 | 4
  Italy | 34 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Phase 2 - Percentage of Participants With Composite Endpoint of Clinical Events
Description: Composite event is defined as the onset of at least one of the following events:
  * supplemental oxygen requirement based on a worsening of PaO2/FiO2 ratio,
  * invasive mechanical ventilation use,
  * admission to Intensive Care Unit (ICU),
  * use of a rescue medication for any reason. Please note that in the measure type "number" actually is a "rate" of patients. Rate is referred to a binomial response rate while the 95% CIs are estimated by using the Clopper-Pearson's method
Time Frame: Up to Day 1
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP. The FAS population was analyzed according to intention to treat (ITT) principle, i.e. by treatment allocation regardless the occurrence of intercurrent events. The FAS population was used for the primary analyses of the study and to present results on efficacy data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
percentage of participants
  Composite event | 16.7 [6.4 to 32.8] | 42.1 [20.3 to 66.5]
  Supplemental oxygen requirement based on PaO2/FiO2 | 13.9 [4.7 to 29.5] | 26.3 [9.1 to 51.2]
  Invasive Mechanical ventilation | 2.8 [0.1 to 14.5] | 5.3 [0.1 to 26.0]
  Admission to ICU | 2.8 [0.1 to 14.5] | 0.0 [0.0 to 17.6]
  Use of a rescue medication for any reason | 0.0 [0.0 to 9.7] | 26.3 [9.1 to 51.2]
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Test type: Superiority; p = 0.02164, Log Rank
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Sensitivity analysis of time to event for each single component of the primary endpoint: Supplemental oxygen requirement based on PaO2/FiO2; Test type: Superiority; p = 0.20043, Log Rank
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Sensitivity analysis of time to event for each single component of the primary endpoint: time to first invasive mechanical ventilation; Test type: Superiority; p = 0.30215, Log Rank
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Sensitivity analysis of time to event for each single component of the primary endpoint: time to first admission to ICU; Test type: Superiority; p = 0.56370, Log Rank
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Sensitivity analysis of time to event for each single component of the primary endpoint: time to first use of a rescue medication for any reason; Test type: Superiority; p = 0.00132, Log Rank

2. Secondary Outcome: Phase 2 - Percentage of Patients With Improvement in Clinical Severity Score (as Recommended by WHO for COVID Studies) of at Least Two Points
Description: Changes in clinical severity score are defined as the time to clinical improvement of two points from the time of randomization on a seven-category ordinal scale or live discharge from the hospital, whichever came first. The seven-category ordinal scale consisted of the following: 1) not hospitalized, with resumption of normal activities; 2) not hospitalized, but unable to resume normal activities; 3) hospitalized, not requiring supplemental oxygen; 4) hospitalized, requiring supplemental oxygen; 5) hospitalized, requiring high-flow oxygen therapy, non-invasive mechanical ventilation, or both; 6) hospitalized, requiring Extracorporeal Membrane Oxygenation (ECMO), invasive mechanical ventilation, or both; and 7) death. The higher the score, the worse the outcome. A subject is considered "improved" with a clinical severity score improvement of at least two points compared to randomization or live discharge from the hospital.
  n are the subjects improved at each time point vs baseline.
Time Frame: At day 1, day 2, week 1, day 21(end of treatment, EOT), EOS (end of study, i.e. 7±3 days after EOT)
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP. The FAS population was analyzed according to intention to treat (ITT) principle, i.e. by treatment allocation regardless the occurrence of intercurrent events. The FAS population was used for the primary analyses of the study and to present results on efficacy data;
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
Percentage of patients
  Day 1: number analyzed (Participants) | 35 | 19
  Day 1 | 0.0 [0.0 to 10.0] | 0.0 [0.0 to 17.6]
  Day 2: number analyzed (Participants) | 35 | 18
  Day 2 | 0.0 [0.0 to 10.0] | 0.0 [0.0 to 18.5]
  Week 1: number analyzed (Participants) | 34 | 17
  Week 1 | 23.5 [10.7 to 41.2] | 17.6 [3.8 to 43.4]
  EOT: number analyzed (Participants) | 34 | 19
  EOT | 26.5 [12.9 to 44.4] | 26.3 [9.1 to 51.2]
  EOS: number analyzed (Participants) | 26 | 9
  EOS | 61.5 [40.6 to 79.8] | 55.6 [21.2 to 86.3]
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); comparison at week 1; Test type: Superiority; p = 0.731, Fisher Exact
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); at EOT; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); at EOS; Test type: Superiority; p = 1.000, Fisher Exact

3. Secondary Outcome: Phase 2 - Percentage of Improved Subjects in Dyspnea Severity, Assessed by Liker Scale
Description: The severity of dyspnea can be measured through the Liker scale. The Liker scale is used as follows: the patient grades his current breathing compared to when he first started the drug (from -3 to 3). "0" = no change, "1" =minimally better, "2" =moderately better, "3" =markedly better, "-1" =minimally worse, "-2" =moderately worse, "-3" =markedly worse. The higher the score, the better the outcome. N is the number of subjects for which the evaluation of the dyspnea severity scale at each time point is available. n is the number of subjects improved at each time point in comparison with the randomization.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment, EOT), 7±3 days after treatment period (end of study, EOS)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
Participants
  Baseline: number analyzed (Participants) | 11 | 6
  Baseline | 0 | 1
  Day 1: number analyzed (Participants) | 16 | 9
  Day 1 | 7 | 2
  Day 2: number analyzed (Participants) | 16 | 7
  Day 2 | 12 | 2
  Week 1: number analyzed (Participants) | 25 | 9
  Week 1 | 23 | 6
  EOT: number analyzed (Participants) | 23 | 9
  EOT | 20 | 6
  EOS: number analyzed (Participants) | 18 | 3
  EOS | 16 | 3
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); at baseline; Test type: Superiority; p = 0.353, Fisher Exact
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); At Day 1; Test type: Superiority; p = 0.401, Fisher Exact
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); At Day 2; Test type: Superiority; p = 0.066, Fisher Exact
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); At week 1; Test type: Superiority; p = 0.102, Fisher Exact
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); at EOT; Test type: Superiority; p = 0.314, Fisher Exact
Statistical Analysis 6: Comparison: Reparixin (FAS) vs Standard of Care (FAS); at EOS; Test type: Superiority; p = 1.000, Fisher Exact

4. Secondary Outcome: Phase 2 - Change From Baseline in Dyspnea Severity, Assessed by VAS Scale
Description: The severity of dyspnea is measured also through the VAS scale. The VAS scale is used as follows: the patient draws a horizontal line on an axial graph (from 0 to 100) to show the degree of how he feels about breathing. The number "0" equals the worst breathing the patient has ever felt and the number "100" equals the best he has ever felt. N is the number of subjects for which the evaluation of the dyspnea severity scale at each time point is available. n is the number of subjects improved at each time point in comparison with the randomization.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment, EOT), 7±3 days after treatment period (end of study, EOS)
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least one dose of the IMP.
  Please note that N (36 for Reparixin and 19 for SoC) is the number of subjects for which the evaluation of the dyspnea severity scale at each time point is available. n - hereunder reported (28 for Reparixin and 19 for SoC) - is the number of subjects improved at each time point in comparison with the randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
score on a scale
  Baseline: number analyzed (Participants) | 8 | 5
  Baseline | 56.9 (37.3) | 4.0 (5.5)
  to Day 1: number analyzed (Participants) | 4 | 4
  to Day 1 | 4.3 (8.5) | 20.0 (40.0)
  to Day 2: number analyzed (Participants) | 4 | 4
  to Day 2 | 32.3 (40.3) | 44.8 (51.7)
  Week 1: number analyzed (Participants) | 5 | 3
  Week 1 | 29.0 (34.0) | 86.0 (5.3)
  EOT: number analyzed (Participants) | 5 | 3
  EOT | 33.0 (41.8) | 89.7 (0.6)
  EOS: number analyzed (Participants) | 2 | 0
  EOS | 22.5 (31.8) |
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1 vs baseline; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change of VAS scale
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2 vs baseline; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change of VAS scale
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); week 1 vs baseline; Test type: Superiority; p = 0.050, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change of VAS scale
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT vs baseline; Test type: Superiority; p = 0.0227, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change of VAS scale

5. Secondary Outcome: Changes From Baseline in Body Temperature to Any Post-baseline Timepoints
Description: Variations in the mean body temperature from baseline to any post-baseline timepoint were assessed.
  n is the number of subjects for which the evaluation of the body temperature at each time point is available.
Time Frame: Baseline, Day 1, Day 2, Week 1, EOT and EOS
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: F°
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
F°
  Baseline | 36.4 (0.5) | 36.5 (0.5)
  to Day 1: number analyzed (Participants) | 34 | 19
  to Day 1 | -0.2 (0.5) | 0.2 (0.9)
  to Day 2: number analyzed (Participants) | 35 | 18
  to Day 2 | -0.1 (0.7) | -0.1 (0.6)
  to Week 1: number analyzed (Participants) | 32 | 14
  to Week 1 | -0.1 (0.6) | -0.2 (0.6)
  to EOT: number analyzed (Participants) | 32 | 15
  to EOT | -0.2 (0.6) | -0.4 (0.6)
  to EOS: number analyzed (Participants) | 10 | 3
  to EOS | -0.1 (0.5) | -0.5 (0.6)
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); At Day 1; Test type: Superiority; p = 0.122, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); At Day 2; Test type: Superiority; p = 0.985, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); at week 1; Test type: Superiority; p = 0.857, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); at EOT; Test type: Superiority; p = 0.436, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); At EOS; Test type: Superiority; p = 0.350, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Phase 2 - Percentage of Subjects Worsened, During Supplemental Oxygen Treatment, From Randomization According to PaO2/FiO2
Description: Cumulative quantity of oxygen treatment (L) = Sum of all Quantity (L) in CONCOMITANT OXYGEN TREATMENT form, from randomization to time point of interest.
  According to PaO2/FiO2, the classification is 'mild' if 200 <= PaO2/FiO2 < 300 mmHg, 'moderate' if 100 <= PaO2/FiO2 < 200 mmHg, 'severe' if PaO2/FiO2 < 100 mmHg. A patient with ARDS (PaO2/FiO2<300 mmHg) is considered 'worsened' in case of a decrease of PaO2/FiO2 of at least one third (-33,3%) from the baseline PaO2/FiO2 value.
  NOTE that: N is the number of subjects for which the evaluation of the PaO2/FiO2 ratio at each time point is available. While n is the number of subjects worsened at each time point in comparison with the randomization, expressed in percentage.
Time Frame: At day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
percentage of subjects
  Day 1 - subjects worsened (%): number analyzed (Participants) | 27 | 14
  Day 1 - subjects worsened (%) | 7.4 [0.9 to 24.3] | 14.3 [1.8 to 42.8]
  Day 2 - subjects worsened (%): number analyzed (Participants) | 31 | 15
  Day 2 - subjects worsened (%) | 12.9 [3.6 to 29.8] | 20.0 [4.3 to 48.1]
  Week 1 - subjects worsened (%): number analyzed (Participants) | 26 | 14
  Week 1 - subjects worsened (%) | 0.0 [0.0 to 13.2] | 21.4 [4.7 to 50.8]
  EOT - subjects worsened (%): number analyzed (Participants) | 29 | 12
  EOT - subjects worsened (%) | 0.0 [0.0 to 11.9] | 8.3 [0.2 to 38.5]
  EOS - subjects worsened (%): number analyzed (Participants) | 10 | 3
  EOS - subjects worsened (%) | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 70.8]
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1; Test type: Superiority — p-values are referred to a two-sided Fisher's Exact test for worsening; p = 0.596, Fisher Exact
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2; Test type: Superiority — p-values are referred to a two-sided Fisher's Exact test for worsening; p = 0.667, Fisher Exact
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1; Test type: Superiority — p-values are referred to a two-sided Fisher's Exact test for worsening; p = 0.037, Fisher Exact
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority — p-values are referred to a two-sided Fisher's Exact test for worsening; p = 0.293, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for worsening

7. Secondary Outcome: Phase 2 - Percentage of Subjects Worsened, During Supplemental Oxygen Treatment, From Randomization According to Oxygen Delivery System Classification
Description: Duration of oxygen administration (hours) = Administration end date/time - Administration start date/time / 60. N is the number of subjects for which the evaluation of the Oxygen Delivery System Classification at each time point is available. n is the number of subjects worsened at each time point, expressed in percentage, in comparison with the randomization. According to Oxygen Delivery System, the classification is 'invasive' if there is Invasive Medicinal Ventilation or ECMO, else 'high flow' if there is High Flow Nasal Cannula or BIPAP or CPAP, else 'low flow' if there is Nasal Cannula or Mask then Class=Low Flow Classification. A patient is considered 'Worsened' after baseline if there is an increase in the level of severity within the oxygen delivery system classification (Invasive > High Flow > Low Flow).
Time Frame: day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
percentage of patients
  Day 1 - subjects worsened | 5.6 [0.7 to 18.7] | 0.0 [0.0 to 17.6]
  Day 2 - subjects worsened | 5.6 [0.7 to 18.7] | 5.3 [0.1 to 26.0]
  Week 1 - subjects worsened: number analyzed (Participants) | 34 | 17
  Week 1 - subjects worsened | 2.9 [0.1 to 15.3] | 17.6 [3.8 to 43.4]
  EOT - subjects worsened: number analyzed (Participants) | 35 | 19
  EOT - subjects worsened | 2.9 [0.1 to 14.9] | 15.8 [3.4 to 39.6]
  EOS - subjects worsened: number analyzed (Participants) | 28 | 12
  EOS - subjects worsened | 3.6 [0.1 to 18.3] | 8.3 [0.2 to 38.5]
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1; Test type: Superiority; p = 0.539, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for worsening and
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for worsening
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1; Test type: Superiority; p = 0.102, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for worsening
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p = 0.119, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for worsening
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS; Test type: Superiority; p = 0.515, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for worsening

8. Secondary Outcome: Phase 2 - Oxygen Cumulative Duration During the Study
Description: This outcome assesses the oxygen cumulative duration during the study. N is the number of subjects for which the evaluation of the PaO2/FiO2 ratio or Oxygen Delivery System Classification at each time point is available. n is the number of subjects worsened at each time point in comparison with the randomization.
Time Frame: Week 1, EOT, EOS
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
hours
  week 1: number analyzed (Participants) | 34 | 18
  week 1 | 141.93 (55.68) | 130.22 (80.89)
  EOT: number analyzed (Participants) | 34 | 18
  EOT | 151.55 (75.53) | 134.00 (86.21)
  EOS: number analyzed (Participants) | 36 | 18
  EOS | 195.26 (198.62) | 155.71 (135.93)
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1; Test type: Superiority; p = 0.366, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for cumulative duration
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p = 0.489, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for cumulative duration
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS; Test type: Superiority; p = 0.486, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for cumulative duration

9. Secondary Outcome: Phase 2 - Oxygen Cumulative Quantity During the Study
Description: In this endpoint is assessed the oxygen cumulative quantity needed at each single timepoint.
  N is the number of subjects for which the evaluation of the PaO2/FiO2 ratio or Oxygen Delivery System Classification at each time point is available. n is the number of subjects worsened at each time point in comparison with the randomization.
Time Frame: Week 1, EOT and EOS
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
liters
  Week 1: number analyzed (Participants) | 33 | 18
  Week 1 | 24.99 (22.22) | 29.20 (29.51)
  EOT: number analyzed (Participants) | 33 | 18
  EOT | 25.64 (22.16) | 29.73 (31.53)
  EOS: number analyzed (Participants) | 35 | 18
  EOS | 26.54 (22.31) | 33.38 (31.64)
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1; Test type: Superiority; p = 0.790, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for cumulative quantity
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p = 0.961, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for cumulative quantity
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS; Test type: Superiority; p = 0.619, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for cumulative quantity

10. Secondary Outcome: Phase 2 - Percentage of Subjects Requiring Mechanical Ventilation Use, Overall
Description: Percentage along with the 95% confidence interval (Clopper-Pearson's formula) of subjects requiring mechanical ventilation are calculated and compared. N is the number of subjects for which the evaluation of the use of mechanical ventilation is available. n is the number, expressed in percentage, of subjects requiring mechanical ventilation, overall.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
percentage of subjects
  Baseline - subjects requiring | 11.1 [3.1 to 26.1] | 10.5 [1.3 to 33.1]
  Day1 - subjects requiring | 11.1 [3.1 to 26.1] | 10.5 [1.3 to 33.1]
  Day 2 - subjects requiring: number analyzed (Participants) | 35 | 18
  Day 2 - subjects requiring | 11.4 [3.2 to 26.7] | 16.7 [3.6 to 41.4]
  Week 1- subjects requiring: number analyzed (Participants) | 34 | 17
  Week 1- subjects requiring | 8.8 [1.9 to 23.7] | 11.8 [1.5 to 36.4]
  EOT - subjects requiring: number analyzed (Participants) | 35 | 19
  EOT - subjects requiring | 8.6 [1.8 to 23.1] | 5.3 [0.1 to 26.0]
  EOS -subjects requiring: number analyzed (Participants) | 27 | 10
  EOS -subjects requiring | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 30.8]
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Baseline; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 3: Comparison: Reparixin (FAS); Day 2; Test type: Superiority; p = 0.678, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 6: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion

11. Secondary Outcome: Phase 2 - Cumulative Duration of Mechanical Ventilation Use, Overall
Description: Cumulative duration of mechanical ventilation (in hours) = Sum of duration of mechanical ventilation (hours) in mechanical ventilation form, from randomization to time point of interest.
  Duration of mechanical ventilation (hours) = End date/time - Start date/time / 60. n is the number of subjects for which the evaluation of the use of mechanical ventilation is available
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
hours
  Week 1: number analyzed (Participants) | 4 | 3
  Week 1 | 162.54 (58.92) | 142.42 (44.89)
  EOT: number analyzed (Participants) | 4 | 3
  EOT | 149.99 (53.23) | 146.86 (43.80)
  EOS: number analyzed (Participants) | 4 | 3
  EOS | 179.51 (78.30) | 154.86 (56.52)
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1; Test type: Superiority; p = 0.696, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for cumulative duration
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney) — p-values are referred to a-sided Wilcoxon test for cumulative duration
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS; Test type: Superiority; p = 0.596, Wilcoxon (Mann-Whitney) — p-values are referred to a-sided Wilcoxon test for cumulative duration

12. Secondary Outcome: Phase 2 - Percentage of Subjects With Intensive Care Unit (ICU) Admission Need
Description: Percentage, along with the 95% confidence interval (Clopper-Pearson's formula), of subjects requiring ICU admission are calculated and compared.N is the number of subjects for which the evaluation of the ICU admission need is available.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
percentage of patients
  Baseline - subjects admitted to ICU | 2.8 [0.1 to 14.5] | 5.3 [0.1 to 26.0]
  Day 1 - subjects admitted to ICU | 2.8 [0.1 to 14.5] | 5.3 [0.1 to 26.0]
  Day 2 - subjects admitted to ICU: number analyzed (Participants) | 35 | 18
  Day 2 - subjects admitted to ICU | 5.7 [0.7 to 19.2] | 5.6 [0.1 to 27.3]
  Week 1 - subjects admitted to ICU: number analyzed (Participants) | 34 | 17
  Week 1 - subjects admitted to ICU | 2.9 [0.1 to 15.3] | 0.0 [0.0 to 19.5]
  EOT - subjects admitted to ICU: number analyzed (Participants) | 35 | 19
  EOT - subjects admitted to ICU | 2.9 [0.1 to 14.9] | 0.0 [0.0 to 17.6]
  EOS - subjects admitted to ICU: number analyzed (Participants) | 27 | 10
  EOS - subjects admitted to ICU | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 12.8]
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Baseline; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1; Test type: Superiority; p = 1.000, Fisher Exact; p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2; Test type: Superiority; p = 1.000, Fisher Exact; p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); week 1; Test type: Superiority; p = 1.000, Fisher Exact; p-values are referred to a two-sided Fisher's Exact test for proportion
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p = 1.000, Fisher Exact — p-values are referred to a two-sided Fisher's Exact test for proportion

13. Secondary Outcome: Phase 2 - Cumulative ICU Stay
Description: Cumulative ICU stay was assessed at different timepoints and measured in days
Time Frame: Day 1, Day 2, Week 1, EOT, EOS
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
days
  Day 1 - cumulative ICU stay: number analyzed (Participants) | 1 | 1
  Day 1 - cumulative ICU stay | 1.0 [1 to 1] | 1.0 [1 to 1]
  Day 2 - cumulative ICU stay: number analyzed (Participants) | 1 | 1
  Day 2 - cumulative ICU stay | 2.0 [2 to 2] | 2.0 [2 to 2]
  Week 1 - cumulative ICU stay: number analyzed (Participants) | 1 | 1
  Week 1 - cumulative ICU stay | 7.0 [7 to 7] | 3.0 [3 to 3]
  EOT - cumulative ICU stay: number analyzed (Participants) | 1 | 1
  EOT - cumulative ICU stay | 6.0 [6 to 6] | 3.0 [3 to 3]
  EOS - cumulative ICU stay: number analyzed (Participants) | 36 | 1
  EOS - cumulative ICU stay | 50.0 [50 to 50] | 3.0 [3 to 3]

14. Secondary Outcome: Phase 2 - Lung Damage Extension by Severity and by Timepoint
Description: Lung damage extensions is assessed by Chest CT or Rx. This damage can be as follows: "none", "trace", "mild", "moderate", or "severe".
  N is the number of subjects for which the evaluation of the lung damage extension at each time point is available.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least one dose of the IMP. Please note that N, hereunder reported, is the number of subjects for which the evaluation of the lung damage extension or lung damage exudation degree at each time point is available (very low at Day 1 and EOS time points in the "Reparixin" Arm and at the Day 1, 2, and Week 1 time points in the "Standard of Care" Arm).
Measure: Number; unit: participants
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
participants
  baseline - none | 0 | 0
  baseline - trace | 1 | 2
  baseline - mild | 9 | 3
  baseline - moderate | 23 | 11
  baseline - severe | 3 | 3
  Day 1 - none: number analyzed (Participants) | 1 | 1
  Day 1 - none | 0 | 0
  Day 1 - trace: number analyzed (Participants) | 1 | 1
  Day 1 - trace | 0 | 0
  Day 1 - mild: number analyzed (Participants) | 1 | 1
  Day 1 - mild | 0 | 1
  Day 1 - moderate: number analyzed (Participants) | 1 | 1
  Day 1 - moderate | 1 | 0
  Day 1 - severe: number analyzed (Participants) | 1 | 1
  Day 1 - severe | 0 | 0
  Day 2 - none: number analyzed (Participants) | 1 | 1
  Day 2 - none | 0 | 0
  Day 2 - trace: number analyzed (Participants) | 1 | 1
  Day 2 - trace | 0 | 0
  Day 2 - mild: number analyzed (Participants) | 1 | 1
  Day 2 - mild | 0 | 1
  Day 2 - moderate: number analyzed (Participants) | 1 | 1
  Day 2 - moderate | 0 | 0
  Day 2 - severe: number analyzed (Participants) | 1 | 1
  Day 2 - severe | 1 | 0
  week 1 - none: number analyzed (Participants) | 12 | 4
  week 1 - none | 0 | 0
  week 1- trace: number analyzed (Participants) | 12 | 4
  week 1- trace | 1 | 0
  week 1 - mild: number analyzed (Participants) | 12 | 4
  week 1 - mild | 6 | 2
  week 1 - moderate: number analyzed (Participants) | 12 | 4
  week 1 - moderate | 4 | 0
  week 1 - severe: number analyzed (Participants) | 12 | 4
  week 1 - severe | 1 | 2
  EOT - none: number analyzed (Participants) | 16 | 19
  EOT - none | 1 | 0
  EOT - trace: number analyzed (Participants) | 16 | 19
  EOT - trace | 3 | 0
  EOT - mild: number analyzed (Participants) | 16 | 19
  EOT - mild | 8 | 2
  EOT - moderate: number analyzed (Participants) | 16 | 19
  EOT - moderate | 3 | 0
  EOT - severe: number analyzed (Participants) | 16 | 19
  EOT - severe | 1 | 2
  EOS - none: number analyzed (Participants) | 2 | 19
  EOS - none | 0 | 0
  EOS - trace: number analyzed (Participants) | 2 | 19
  EOS - trace | 0 | 0
  EOS - mild: number analyzed (Participants) | 2 | 19
  EOS - mild | 1 | 1
  EOS - moderate: number analyzed (Participants) | 2 | 19
  EOS - moderate | 1 | 1
  EOS - severe: number analyzed (Participants) | 2 | 19
  EOS - severe | 0 | 0
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); baseline; Test type: Superiority; p = 0.760, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1; Test type: Superiority; p = 0.394, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p = 0.141, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test

15. Secondary Outcome: Phase 2 - Lung Exudation by Severity and by Timepoint
Description: Lung exudation is assessed by Chest CT or Rx. This can be as follows: "none", "trace", "mild", "moderate", or "severe".
  N is the number of subjects for which the evaluation of the lung damage extension at each time point is available.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
participants
  baseline - none | 32 | 18
  baseline - trace | 0 | 0
  baseline - mild | 1 | 0
  baseline - moderate | 3 | 1
  baseline - severe | 0 | 0
  Day 1 - none: number analyzed (Participants) | 1 | 1
  Day 1 - none | 0 | 0
  Day 1 - trace: number analyzed (Participants) | 1 | 1
  Day 1 - trace | 0 | 0
  Day 1 - mild: number analyzed (Participants) | 1 | 1
  Day 1 - mild | 0 | 0
  Day 1 - moderate: number analyzed (Participants) | 1 | 1
  Day 1 - moderate | 1 | 1
  Day 1 - severe: number analyzed (Participants) | 1 | 1
  Day 1 - severe | 0 | 0
  Day 2 - none: number analyzed (Participants) | 1 | 1
  Day 2 - none | 0 | 0
  Day 2 - trace: number analyzed (Participants) | 1 | 1
  Day 2 - trace | 0 | 0
  Day 2 - mild: number analyzed (Participants) | 1 | 1
  Day 2 - mild | 0 | 1
  Day 2 - moderate: number analyzed (Participants) | 1 | 1
  Day 2 - moderate | 0 | 0
  Day 2 - severe: number analyzed (Participants) | 1 | 1
  Day 2 - severe | 1 | 0
  week 1 - none: number analyzed (Participants) | 12 | 4
  week 1 - none | 12 | 3
  week 1- trace: number analyzed (Participants) | 12 | 4
  week 1- trace | 0 | 0
  week 1 - mild: number analyzed (Participants) | 12 | 4
  week 1 - mild | 0 | 0
  week 1 - moderate: number analyzed (Participants) | 12 | 4
  week 1 - moderate | 0 | 0
  week 1 - severe: number analyzed (Participants) | 36 | 4
  week 1 - severe | 12 | 1
  EOT - none: number analyzed (Participants) | 16 | 4
  EOT - none | 15 | 3
  EOT - trace: number analyzed (Participants) | 16 | 4
  EOT - trace | 0 | 0
  EOT - mild: number analyzed (Participants) | 16 | 4
  EOT - mild | 1 | 0
  EOT - moderate: number analyzed (Participants) | 16 | 19
  EOT - moderate | 0 | 4
  EOT - severe: number analyzed (Participants) | 16 | 4
  EOT - severe | 0 | 0
  EOS - none: number analyzed (Participants) | 2 | 2
  EOS - none | 2 | 2
  EOS - trace: number analyzed (Participants) | 2 | 2
  EOS - trace | 0 | 0
  EOS - mild: number analyzed (Participants) | 2 | 2
  EOS - mild | 0 | 0
  EOS - moderate: number analyzed (Participants) | 2 | 2
  EOS - moderate | 0 | 0
  EOS - severe: number analyzed (Participants) | 2 | 2
  EOS - severe | 0 | 0
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); baseline; Test type: Superiority; p = 0.500, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); week 1; Test type: Superiority; p = 0.112, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT; Test type: Superiority; p = 0.277, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test

16. Secondary Outcome: Phase 2 - Change From Baseline in Partial Arterial Oxygen Pressure (PaO2)
Description: PaO2 measures the pressure of oxygen dissolved in the blood and how well oxygen is able to move from the airspace of the lungs into the blood.
  Normally, PaO2 is between 75 and 100 mmHg (at sea level). Lower levels indicate an unsufficient amount of oxygen flowing from the alveoli to the blood. Please note that a significant proportion of patients in both groups did not have post-baseline assessments of PaO2.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least one dose of the IMP. Please note that N, hereunder reported, is the number of subjects for which the evaluation of the PaO2 at each time point is available (very low at Day 1 and EOS time points in the "Reparixin" Arm and at the Day 1, 2, and Week 1 time points in the "Standard of Care" Arm).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
mmHg
  Baseline: number analyzed (Participants) | 17 | 8
  Baseline | 121.69 (47.15) | 68.64 (9.23)
  to Day 1: number analyzed (Participants) | 8 | 4
  to Day 1 | -19.61 (50.09) | 14.20 (25.76)
  to Day 2: number analyzed (Participants) | 13 | 4
  to Day 2 | 12.62 (60.20) | -4.68 (14.03)
  to week 1: number analyzed (Participants) | 10 | 3
  to week 1 | 11.76 (25.26) | -1.13 (54.80)
  to EOT: number analyzed (Participants) | 11 | 1
  to EOT | 8.01 (36.08) | -18.70
  to EOS: number analyzed (Participants) | 8 | 1
  to EOS | -35.76 (47.84) | 1.80
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1 vs baseline; Test type: Superiority; p = 0.2027, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2 vs baseline; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Week 1 vs baseline; Test type: Superiority; p = 0.4469, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT vs baseline; Test type: Superiority; p = 0.2466, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS vs baseline; Test type: Superiority; p = 0.1752, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change

17. Secondary Outcome: Phase 2 - Change From Baseline in Oxygen Saturation (SpO2)
Description: SpO2 measures the amount of oxygen-carrying hemoglobin in the blood relative to the amount of hemoglobin not carrying oxygen. Acceptable normal ranges for patients without pulmonary pathology are from 95 to 99 percent.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent of oxygen saturation
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
percent of oxygen saturation
  Baseline: number analyzed (Participants) | 35 | 18
  Baseline | 95.79 (3.17) | 94.97 (2.60)
  to Day 1: number analyzed (Participants) | 29 | 18
  to Day 1 | 0.17 (2.20) | -0.41 (3.57)
  to Day 2: number analyzed (Participants) | 32 | 17
  to Day 2 | 0.38 (2.88) | -0.63 (3.86)
  to week 1: number analyzed (Participants) | 30 | 13
  to week 1 | 1.18 (3.34) | 0.73 (3.71)
  to EOT: number analyzed (Participants) | 29 | 14
  to EOT | 0.88 (3.57) | 1.19 (3.89)
  to EOS: number analyzed (Participants) | 10 | 2
  to EOS | 0.47 (3.17) | -4.00 (1.41)
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1 vs baseline; Test type: Superiority; p = 0.6441, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2 vs baseline; Test type: Superiority; p = 0.3529, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); week 1 vs baseline; Test type: Superiority; p = 0.3581, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT vs baseline; Test type: Superiority; p = 0.1666, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS vs baseline; Test type: Superiority; p = 0.0851, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change

18. Secondary Outcome: Phase 2 - Partial Arterial Oxygen Pressure (PaO2) to Fraction of Inspiration O2 (FiO2) Ratio [PaO2/FiO2 Ratio]
Description: PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage) also known as the Horowitz index, the Carrico index, and (most conveniently) the P/F ratio at sea level, the normal PaO2/FiO2 ratio is ~ 400-500 mmHg (~55-65 kPa).
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
ratio
  Baseline: number analyzed (Participants) | 34 | 17
  Baseline | 186.82 (64.86) | 196.91 (58.49)
  To day 1: number analyzed (Participants) | 27 | 14
  To day 1 | 21.58 (65.81) | 6.08 (125.00)
  To day 2: number analyzed (Participants) | 31 | 15
  To day 2 | 48.29 (154.49) | -8.53 (71.74)
  To week 1: number analyzed (Participants) | 26 | 14
  To week 1 | 160.80 (137.83) | 54.28 (138.36)
  To EOT: number analyzed (Participants) | 29 | 12
  To EOT | 171.27 (149.56) | 74.65 (113.55)
  To EOS: number analyzed (Participants) | 10 | 3
  To EOS | 199.26 (85.45) | 84.87 (67.92)
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1 vs baseline; Test type: Superiority; p = 0.3359, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2 vs baseline; Test type: Superiority; p = 0.3136, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); week 1 vs baseline; Test type: Superiority; p = 0.0441, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT vs baseline; Test type: Superiority; p = 0.0965, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS vs baseline; Test type: Superiority; p = 0.0519, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change

19. Secondary Outcome: Phase 2 - Change From Baseline in Reactive Protein (CRP)
Description: For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L). Levels between 10 mg/L and 100 mg/L are moderately elevated and are usually due to more significant inflammation from an infectious or non-infectious cause. Inflammatory status is documented by C-reactive protein (CRP) ≥ 100mg/L.
Time Frame: Baseline, day 1, day 2, week 1, day 21(end of treatment), follow-up (FU) (7±3 days after treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Reparixin (FAS) | Standard of Care (FAS)
Number analyzed (Participants) | 36 | 19
mg/L
  baseline: number analyzed (Participants) | 35 | 19
  baseline | 57.04 (41.44) | 58.87 (57.25)
  to day 1: number analyzed (Participants) | 11 | 9
  to day 1 | -0.14 (73.28) | 38.46 (117.19)
  to day 2: number analyzed (Participants) | 22 | 8
  to day 2 | -29.24 (37.66) | -2.15 (52.37)
  to week 1: number analyzed (Participants) | 26 | 14
  to week 1 | -39.09 (56.56) | 0.52 (80.24)
  to EOT: number analyzed (Participants) | 24 | 13
  to EOT | -40.88 (50.27) | -25.28 (87.16)
  to EOS: number analyzed (Participants) | 11 | 7
  to EOS | -49.43 (57.65) | -45.20 (78.97)
Statistical Analysis 1: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 1 vs baseline; Test type: Superiority; p = 0.470, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 2: Comparison: Reparixin (FAS) vs Standard of Care (FAS); Day 2 vs baseline; Test type: Superiority; p = 0.425, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 3: Comparison: Reparixin (FAS) vs Standard of Care (FAS); week 1 vs baseline; Test type: Superiority; p = 0.086, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 4: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOT vs baseline; Test type: Superiority; p = 0.600, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change
Statistical Analysis 5: Comparison: Reparixin (FAS) vs Standard of Care (FAS); EOS vs baseline; Test type: Superiority; p = 0.717, Wilcoxon (Mann-Whitney) — p-values are referred to a two-sided Wilcoxon test for differences in the change

ADVERSE EVENTS:
Time Frame: Throughout the study, till day 21
Description: The Safety set (SAF), which consisted of all randomized subjects who received at least one dose of the investigational medicinal product (IMP).
Groups:
- Reparixin (SAF): Reparixin was administered via oral tablets 1200 mg TID for 7 days. In case of improvement, treatment can be prolonged at discretion of the investigator up to a maximum of 21 days of treatment in total or live discharge from the hospital, whichever comes first.
- Standard of Care (SAF): Standard of care, which is defined as any drug currently used to treat the COVID-19 pneumonia.
Arm/Group | Reparixin (SAF) | Standard of Care (SAF)
All-Cause Mortality (participants affected / at risk) | 1/36 | 3/19
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/19
Other Adverse Events (participants affected / at risk) | 1/36 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin (SAF) (N=36) | Standard of Care (SAF) (N=19)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin (SAF) (N=36) | Standard of Care (SAF) (N=19)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT04794803/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT04794803/SAP_001.pdf